CLINICAL TRIAL: NCT07117318
Title: Rectal Non-steroid Anti-inflammatory Drugs With or Without Prophylactic Pancreatic Duct Stent for Prevention of Post-ERCP Pancreatitis: a Multicenter, Randomized, Non-inferiority Trial
Brief Title: Rectal NSAIDs With/Without PD Stent for PEP Prevention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, Professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: KY20252177-F-1
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Post-ERCP Acute Pancreatitis; Non-steroid Anti-inflammatory Drugs; Pancreatic Duct Stent Placement
MeSH Terms: interventions — Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NSAIDs alone (Experimental): All patients without contraindications should receive 100mg rectal indomethacin or diclofenac within 30mins before ERCP procedure
  Interventions: Drug: NSAIDs
- NSAIDs plus PDS (Active Comparator): All patients without contraindications should receive 100mg rectal indomethacin or diclofenac within 30mins before ERCP procedure. When eligibility is met, PDS placement will be performed by ERCP colonoscopists.
  Interventions: Device: NSAIDs plus PDS

INTERVENTIONS:
Drug: NSAIDs — All patients without contraindications should receive 100mg rectal indomethacin or diclofenac within 30mins before ERCP procedure
  Arms: NSAIDs alone
Device: NSAIDs plus PDS — All patients without contraindications should receive 100mg rectal indomethacin or diclofenac within 30mins before ERCP procedure. When eligibility is met, PDS placement will be performed by ERCP colonoscopists.
  Arms: NSAIDs plus PDS

SUMMARY:
Pancreatitis is the most common and serious complication following post-endoscopic retrograde cholangiopancreatography (ERCP) and is associated with occasional mortality, extended hospital stays, and increased healthcare expenses. Rectal non-steroidal anti-inflammatory drugs (NSAIDs) and pancreatic duct stent (PDS) placement were demonstrated to be effective strategyies to reduce PEP incidences, particlularly in high-risk patients for post-ERCP pancreatitis (PEP).

Rectal NSAIDs were easy-to-use and safe, while PDS placement were technically complex and carried higher risks of adverse events. A previous network meta-analysis suggested rectal NSAIDs in combination with PDS placement did not differ from rectal NSAIDs alone in PEP prevention. To invesigate if rectal NSAIDs alone could obivate the need of PDS placement, a recent trial from Elmunzer et al. conducted a randomized trial to investigate if rectal NSAIDs alone was non-inferior to the combination of NSAIDs with PDS in high-risk patients. The trial found that the PEP incidence rate in combination group was significantly lower than that in NSAIDs alone group. However, post-hoc analysis of the study suggested that the combination strategy conferred significant benefits only in high-risk patients with pancreatic duct (PD) wire passage, but not in those with other risk factors. Therefore, we hypothesized that rectal NSAIDs alone may obivate the need of PDS in high-risk patients without PD wire passages. Here, we conducted a multicenter, randomized and non-inferiority trial to investigate whether rectal NSAIDs alone is non-inferior to NSAIDs plus PDS placement in high-risk patients without PD wire passages.

ELIGIBILITY:
Inclusion Criteria:

* 18-90 years old patients with native papilla who planned to undergo ERCP
* high-risk patients for post-ERCP pancreatitis must meet one or more following criteria: clinical suspicion of sphincter of Oddi dysfunction, a history of PEP, pancreatic sphincterotomy, precut sphincterotomy, difficult cannulation (>5 cannulation attempts, or >5mins cannulation time, or >1 unintentional pancreatic duct cannulation), or ballon dilatation of an intact biliary sphincter ≤ 1 min, double-wire cannulation. Additionally, patients were considered high-risk if they fulfilled two or more of the following minor criteria: female gender under 50 years old, a history of recurrent pancreatitis (two or more episodes), three or more contrast injections into the pancreatic duct with at least one injection reaching the tail of the pancreas, opacification of pancreatic acini, or brush cytology performed on the pancreatic duct.

Exclusion Criteria:

* Previous biliary sphincterotomy and papillary large balloon dilation
* Planned for placements of pancreatic duct stents (eg. pancreatic duct strictures, planned ampullectomy)
* Allergy to NSAIDs
* The administration of NSAIDs within 7 days
* Not suitable for NSAIDs administration (gastrointestinal hemorrhage within 4 weeks, renal dysfunction [Cr >1.4mg/dl=120umol/l]; presence of coagulopathy before the procedure)
* Acute pancreatitis within 7 days before ERCP or acute pancreatitis with obvious Pancreatic edema and peripancreatic fluid collections
* Hemodynamical instability
* Pregnancy or lactation
* high-risk patients with pancreatic duct wire passages

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1278 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Rate of post-ERCP Pancreatitis | 30 days
  a new or aggravated upper abdominal pain, with an elevated pancreatic enzyme of at least 3 times as the upper limit of normal value 24h after procedure and prolonged hospitalization days for at least 2 days. This definition was based on a widely recognized Cotton consensus

SECONDARY OUTCOMES:
Rate of mild, moderate or severe PEP | 30 days
  The severity classification of post-ERCP pancreatitis was defined according to the Cotton Criteria. Mild PEP: with an extension of hospitalization period of 2-3 days; Moderate PEP: with an extension of hospitalization period of 4-10 days; Severe PEP: with an extension of more than 10 days, or hemorrhagic pancreatitis, phlegmon, or pseudocyst, intervention (percutaneous drainage or surgery), or death.
Rate of patients with different severity of pancreatitis evaluated by revised Atlanta criteria | 30 days
  Mild: The most common form of acute pancreatitis, without organ failure or local or systemic complications, generally resolving within 1 week of onset. Moderately Severe: the presence of transient organ failure, local complications or exacerbation of co-morbid disease.
  Severe: persistent organ failure, that is, organ failure >48 h. Local complications are peripancreatic fluid collections, pancreatic and peripancreatic necrosis (sterile or infected), pseudocyst and walled-off necrosis (sterile or infected).
Rate of ERCP-related perforation | 30 days
  Perforation was established according to Cotton criteria, Mild: slight leakage of fluid or contrast dye, manageable through fluid administration and suction therapy ≤3 days Moderate: definite perforation required to be managed for 4-10 days Severe: management for more than 10 days or requiring for percutaneous or surgical intervention.
Rate of ERCP-related infection | 30 days
  Infection was established according to Cotton criteria. Mild: temperature >38# for 24-48h Moderate: Febrile illness requiring >3 days of hospital treatment; endoscopic or percutaneous interventions; Severe: septic shock or requiring surgery.
Rate of ERCP-related bleeding | 30 days
  Bleeding was established according to Cotton criteria. Mild: a documented decrease in hemoglobin concentration by <3 g/L, without requiring the blood transfusion; Moderate: blood transfusion ≤4 units; without need for angiographic or surgery interventions Severe: Transfusion: ≥5 units or requiring for angiographic or surgery interventions.
The rate of total adverse events | 30 days
  Adverse events include ERCP-related or non ERCP-related adverse events
The rate of successful pancreatic duct stent placements | 1 day

CONTACTS AND LOCATIONS:
Locations (15):
- China (15):
  - The first medical center, Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Department of gastroenterology, Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Department of Gastroenterology, Fujian Medical University Xiamen Humanity Hospital, Xiamen, Fujian
  - Harbin Medical University Affiliated Fourth Hospital, Harbin, Heilongjiang
  - The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Department of Gastroenterology, Huaihe Hospital of Henan University, Kaifeng, Henan
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - 986 Hospital of Xijing Hospital, Xi'an, Shaanxi
  - Xijing of Digestive Diseases, Xi'an, Shaanxi
  - Department of Gastroenterology, The 960th Hospital of the PLA, Jinan, Shandong
  - Shandong Provincial Third Hospital, Jinan, Shandong
  - Department of Endoscopy, Eastern Hepatobiliary Hospital, Second Military Medical University, Shanghai, Shanghai Municipality
  - Affiliated Hangzhou First People's Hospital, Hangzhou, Zhejiang
  - the First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dumonceau JM, Kapral C, Aabakken L, Papanikolaou IS, Tringali A, Vanbiervliet G, Beyna T, Dinis-Ribeiro M, Hritz I, Mariani A, Paspatis G, Radaelli F, Lakhtakia S, Veitch AM, van Hooft JE. ERCP-related adverse events: European Society of Gastrointestinal Endoscopy (ESGE) Guideline. Endoscopy. 2020 Feb;52(2):127-149. doi: 10.1055/a-1075-4080. Epub 2019 Dec 20. PMID 31863440
- [Background] Elmunzer BJ, Foster LD, Serrano J, Cote GA, Edmundowicz SA, Wani S, Shah R, Bang JY, Varadarajulu S, Singh VK, Khashab M, Kwon RS, Scheiman JM, Willingham FF, Keilin SA, Papachristou GI, Chak A, Slivka A, Mullady D, Kushnir V, Buxbaum J, Keswani R, Gardner TB, Forbes N, Rastogi A, Ross A, Law J, Yachimski P, Chen YI, Barkun A, Smith ZL, Petersen B, Wang AY, Saltzman JR, Spitzer RL, Ordiah C, Spino C, Durkalski-Mauldin V; SVI Study Group. Indomethacin with or without prophylactic pancreatic stent placement to prevent pancreatitis after ERCP: a randomised non-inferiority trial. Lancet. 2024 Feb 3;403(10425):450-458. doi: 10.1016/S0140-6736(23)02356-5. Epub 2024 Jan 11. PMID 38219767
- [Background] Han S, Zhang J, Durkalski-Mauldin V, Foster LD, Serrano J, Cote GA, Bang JY, Varadarajulu S, Singh VK, Khashab M, Kwon RS, Scheiman JM, Willingham FF, Keilin SA, Groce JR, Lee PJ, Krishna SG, Chak A, Slivka A, Mullady D, Kushnir V, Buxbaum J, Keswani R, Gardner TB, Wani S, Edmundowicz SA, Shah RJ, Forbes N, Rastogi A, Ross A, Law J, Yachimski P, Chen YI, Barkun A, Smith ZL, Petersen BT, Wang AY, Saltzman JR, Spitzer RL, Spino C, Elmunzer BJ, Papachristou GI; SVI Study Group. Impact of difficult biliary cannulation on post-ERCP pancreatitis: secondary analysis of the stent versus indomethacin trial dataset. Gastrointest Endosc. 2025 Mar;101(3):617-628. doi: 10.1016/j.gie.2024.10.003. Epub 2024 Oct 9. PMID 39389431
- [Background] Akbar A, Abu Dayyeh BK, Baron TH, Wang Z, Altayar O, Murad MH. Rectal nonsteroidal anti-inflammatory drugs are superior to pancreatic duct stents in preventing pancreatitis after endoscopic retrograde cholangiopancreatography: a network meta-analysis. Clin Gastroenterol Hepatol. 2013 Jul;11(7):778-83. doi: 10.1016/j.cgh.2012.12.043. Epub 2013 Jan 30. PMID 23376320
- [Background] Halttunen J, Keranen I, Udd M, Kylanpaa L. Pancreatic sphincterotomy versus needle knife precut in difficult biliary cannulation. Surg Endosc. 2009 Apr;23(4):745-9. doi: 10.1007/s00464-008-0056-0. Epub 2008 Jul 23. PMID 18649101